CLINICAL TRIAL: NCT03857529
Title: Contralaterally Controlled FES Plus Transcranial Direct Current Stimulation for Hand Motor Control After Stroke: A Pilot Study
Brief Title: Improving Stroke Motor Control With Non-invasive Brain Stimulation and Functional Electrical Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, David Cunningham, Assistant Professor, Physical Medicine and Rehabilitation, School of Medicine, MetroHealth Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB18-00197
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Rehabilitation; Hand
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- conventional tDCS concurrent with CCFES (Experimental): tDCS anode placed over the lesioned hemisphere and cathode placed over the non-lesioned hemisphere
  Interventions: Device: transcranial direct current stimulation and electrical stimulator
- unconventional tDCS concurrent with CCFES (Experimental): tDCS cathode placed over the lesioned hemisphere and anode placed over the non-lesioned hemisphere
  Interventions: Device: transcranial direct current stimulation and electrical stimulator
- conventional tDCS preceding CCFES (Experimental): tDCS anode placed over the lesioned hemisphere and cathode placed over the non-lesioned hemisphere
  Interventions: Device: transcranial direct current stimulation and electrical stimulator
- unconventional tDCS preceding CCFES (Experimental): tDCS cathode placed over the lesioned hemisphere and anode placed over the non-lesioned hemisphere
  Interventions: Device: transcranial direct current stimulation and electrical stimulator
- sham tDCS with CCFES (Sham Comparator): sham tDCS preceding and concurrent with CCFES
  Interventions: Device: transcranial direct current stimulation and electrical stimulator

INTERVENTIONS:
Device: transcranial direct current stimulation and electrical stimulator — Contralaterally Controlled Functional Electrical Stimulation: An electrical stimulator will be used to deliver electrical current through surface electrodes to produce hand opening by making the paretic finger and thumb extensor muscles contract. The stimulator will be programmed to deliver stimulation with an intensity that corresponds to the opening of a glove instrumented with sensors and plugged into the stimulator (i.e., CCFES).
  Transcranial direct current stimulation (tDCS): TDCS is a method of noninvasive stimulation of the brain. Using electrodes placed in saline-soaked sponges, low level of direct current (1mA) is delivered over the scalp. This intervention is considered safe and noninvasive because it does not involve implantation or injection or any skin penetration.

SUMMARY:
This pilot study for stroke patients with chronic upper limb hemiplegia will examine the effects of non-invasive brain stimulation and neuromuscular electrical stimulation on hand motor control and corticospinal excitability. Specifically, this study will investigate the effects of timing and delivery of tDCS in conjunction with contralaterally controlled functional electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21
2. ≥ 6 months since first clinical hemorrhagic or nonhemorrhagic stroke
3. Able to follow 3-stage commands and remember 2 of 3 items after 30 minutes
4. Full volitional elbow extension/flexion and hand opening/closing of unaffected limb
5. Adequate active movement of shoulder and elbow to position the paretic hand in the workspace for table-top task practice
6. Patient must be able to sit unassisted in an armless straight-back chair for the duration of the screening portion of the eligibility assessment
7. Medically stable
8. ≥ 10° finger extension
9. Unilateral upper limb hemiparesis with finger extensor strength of ≤ grade 4/5 on the manual muscle test AND a score of

   ≥1 and ≤ 11/14 on the hand section of the upper extremity Fugl-Meyer Assessment
10. Skin intact on hemiparetic arm, hand and scalp
11. While relaxed, surface neuromuscular electrical stimulation of finger extensors and thumb extensors and/or abductors produces a functional degree of hand opening without pain.
12. No significant visual or hearing impairment

Exclusion Criteria:

1. Co-existing neurological condition other than prior stroke involving the hemiparetic upper limb (e.g., peripheral nerve injury, Parkinson's disease, spinal cord injury, traumatic brain injury, multiple sclerosis).
2. Uncontrolled seizure disorder
3. Use of seizure lowering threshold medications at the discretion of the study physician (Dr. Rich Wilson)
4. Cardiac pacemaker or other implanted electronic device and/or stent
5. Pregnant
6. Intramuscular botox injections in any upper extremity muscle in the last 3 months
7. Insensate arm, forearm, or hand
8. Severely impaired cognition and communication
9. Uncompensated hemi-neglect (extinguishing to double simultaneous stimulation)
10. Severe shoulder or hand pain (unable to position hand in the workspace without pain)
11. Metal implant in the head

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Corticospinal Excitability | up to one hour post intervention
  Change in corticospinal excitability will be measured with transcranial magnetic stimulation
Reaction Time | up to one hour post intervention
  Change in reaction time will be assessed with visual and auditory cues.

CONTACTS AND LOCATIONS:
Overall Officials: David A Cunningham, PhD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and results will be made available by request